CLINICAL TRIAL: NCT01966874
Title: Mifepristone and Misoprostol for the Termination of Pregnancy up to 70 Days Gestation
Status: Completed | Type: Observational
Sponsor: Gynuity Health Projects (Other)
Collaborators: Secretaria de Salud, Mexico (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1002
Record Dates: First submitted 2013-10-16; First posted 2013-10-22 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Medical; Abortion, Fetus
Keywords: Medical abortion; Mifepristone; Misoprostol; Zacafemyl; Mexico

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Study population: All study participants will receive 200 mg of the mifepristone product "Zacafemyl", followed 24-48 hours later by 800 mcg of misoprostol.

SUMMARY:
The purpose of this study is to determine the efficacy and acceptability of a regimen of 200 mg mifepristone (Zacafemyl), followed 24-48 hours later by 800 mcg of buccal misoprostol.

DETAILED DESCRIPTION:
In Mexico City, the registration of a new mifepristone product signals a new wave in the SSDF's program for terminating pregnancies up to 70 days. This study evaluates the efficacy of the product Zacafemyl for the termination of pregnancy up to 70 days LMP. It also evaluates the incidence and acceptability of side effects of the medication and regimen. Participants are women of reproductive age with a gestational age of less than or equal to 70 days who want and are eligible for medical abortion, are willing and able to provide all follow up information, and have no contraindications.

Women who are eligible and consent to enroll in the study will be given 200 mg of mifepristone orally in the clinic. The participants will then be given 800 mcg of misoprostol (four 200 mcg tablets) to take home and instructed to take two tablets bucally 24-48 hours after the mifepristone and the remaining tablets within 30 minutes. They will be warned of the side effects they may experience.

All participants will be informed that they can call the clinic in case they have questions about the symptoms or side effects or if they have other concerns. They will also be told that they can return to the clinic in case of severe or persistent bleeding, or if they decide at any point that they want surgical intervention. Participants will also be informed as to the signs of pregnancy termination.

Seven days after taking the mifepristone (the eighth day of the study) the woman should return to the clinic for follow up. Information will be collected on a series of six semi-structured forms that are filled out by members of the study team in accordance with the responses of the participants to the interview questions and the results of physical exams, ultrasounds, etc. Analyses of the data will focus on efficacy, acceptability, side effects, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Women of reproductive age
* Gestational age less than or equal to 70 days LMP
* Willing and capable of accepting and participating
* Eligible for medical abortion according to the clinic's evaluation
* Willing to undergo a surgical intervention to complete the abortion if necessary
* Willing to provide an address and/or telephone number for follow up
* Have easy, straightforward access to a telephone and emergency transport

Exclusion Criteria:

* Gestational age is greater than 70 days LMP
* Suspicion or diagnosis of ectopic pregnancy or undiagnosed adnexal mass
* Use of IUD (note: the woman will be eligible when she removes the IUD)
* Chronic renal failure
* Current long term treatment with corticosteroids
* Allergy to mifepristone, misoprostol, or other prostaglandin
* Coagulopathies or current treatment with anti-coagulants
* Hereditary porphyrias

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women at the study clinics who want medical abortion and meet eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1001 (Actual)
Dates: Start 2011-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Efficacy | One week after enrollment
  Was the method effective in terminating pregnancy? This will be determined by the need for surgical intervention and the dose of misoprostol required.

SECONDARY OUTCOMES:
Acceptability | One week after enrollment
  Was the method acceptable from the perspective of the woman? Were the side effects acceptable to women? Was the buccal route acceptable to women? Responses will be marked as "very satisfied", "satisfied", "neither satisfied nor unsatisfied", "unsatisfied", or "very unsatisfied".

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, Principal Investigator — Gynuity Health Projects; Patricio Sanhueza Smith, Principal Investigator — Secretaria de Salud, Mexico; Maria Laura Garcia, Principal Investigator — M.I. Inguaran; Ana Gabriela Arangure Peraza, Principal Investigator — C.S. Beatriz Velasco
Locations (1):
- Gynuity Health Projects, New York, New York, United States

REFERENCES:
- [Background] Grupo de Informacion en Reproduccion Elegida (GIRE). El aborto en los codigos penales de las entidades federativas. Citacion obtenida por Internet el 8 de octubre de 2007. http://www.gire.org.mx/contenido.php?informacion=31
- [Background] Bracken H, Ngoc NT, Schaff E, Coyaji K, Ambardekar S, Westheimer E, Winikoff B. Mifepristone followed in 24 hours to 48 hours by misoprostol for late first-trimester abortion. Obstet Gynecol. 2007 Apr;109(4):895-901. doi: 10.1097/01.AOG.0000259319.18958.76. PMID 17400851
- [Background] Ashok PW, Hamoda H, Flett GM, Kidd A, Fitzmaurice A, Templeton A. Patient preference in a randomized study comparing medical and surgical abortion at 10-13 weeks gestation. Contraception. 2005 Feb;71(2):143-8. doi: 10.1016/j.contraception.2004.08.013. PMID 15707565
- [Background] Ashok PW, Kidd A, Flett GM, Fitzmaurice A, Graham W, Templeton A. A randomized comparison of medical abortion and surgical vacuum aspiration at 10-13 weeks gestation. Hum Reprod. 2002 Jan;17(1):92-8. doi: 10.1093/humrep/17.1.92. PMID 11756368
- [Background] Gouk EV, Lincoln K, Khair A, Haslock J, Knight J, Cruickshank DJ. Medical termination of pregnancy at 63 to 83 days gestation. Br J Obstet Gynaecol. 1999 Jun;106(6):535-9. doi: 10.1111/j.1471-0528.1999.tb08320.x. PMID 10426609
- [Background] Hamoda H, Ashok PW, Flett GM, Templeton A. A randomised controlled trial of mifepristone in combination with misoprostol administered sublingually or vaginally for medical abortion up to 13 weeks of gestation. BJOG. 2005 Aug;112(8):1102-8. doi: 10.1111/j.1471-0528.2005.00638.x. PMID 16045525
- [Background] Hamoda H, Ashok PW, Flett GM, Templeton A. A randomized trial of mifepristone in combination with misoprostol administered sublingually or vaginally for medical abortion at 13-20 weeks gestation. Hum Reprod. 2005 Aug;20(8):2348-54. doi: 10.1093/humrep/dei037. Epub 2005 May 5. PMID 15878927
- [Background] Hamoda H, Ashok PW, Flett GM, Templeton A. Medical abortion at 9-13 weeks' gestation: a review of 1076 consecutive cases. Contraception. 2005 May;71(5):327-32. doi: 10.1016/j.contraception.2004.10.015. PMID 15854631
- [Background] Datos no publicados. Comunicacion personal I. Dzuba, Gynuity Health Projects, 22 de junio del 2011.
- [Background] Winikoff B, Dzuba IG, Creinin MD, Crowden WA, Goldberg AB, Gonzales J, Howe M, Moskowitz J, Prine L, Shannon CS. Two distinct oral routes of misoprostol in mifepristone medical abortion: a randomized controlled trial. Obstet Gynecol. 2008 Dec;112(6):1303-1310. doi: 10.1097/AOG.0b013e31818d8eb4. PMID 19037040